CLINICAL TRIAL: NCT00592059
Title: A Phase II Study of Systemic Consolidation Therapy With Paclitaxel Plus Carboplatin Following Radical Hysterectomy and Adjuvant Chemoradiation for High Risk Early Stage Cervical Cancer
Brief Title: Systemic Consolidation Therapy After Chemoradiation Therapy Following Operation for High Risk Early Stage Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae Weon Kim, Seoul National University Hospital
Other Study IDs: Sece-1
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the therapeutic efficacy and complications of systemic consolidation therapy with paclitaxel plus carboplatin following radical hysterectomy and adjuvant chemoradiation for high risk early stage cervical cancer.

DETAILED DESCRIPTION:
Systemic consolidation therapy with paclitaxel plus carboplatin (3 cycles per 3 weeks) following radical hysterectomy and adjuvant chemoradiation (3 cycles per 3 weeks) for high risk early stage cervical cancer will elevate the therapeutic efficacy by removing the microscopic metastatic lesions which could not be identified by naked eye and diagnostic imaging tests.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent radical hysterectomy for cervical cancer stage IB-IIA
* Patients who had at least one of the following risk factors in pathologic results; lymph node metastasis, positive residual resection margin, parametrial invasion
* above 20 years
* GOG performance status 0-2
* Informed consent
* Platelet>100K, Hb> 10.0 g/dl, ANC>1500/mm3, Cr <1.25*upper normal limit, bilirubin<1.5mg/dl, AST & ALT<*3 upper normal limit
* Expected life > 6 months

Exclusion Criteria:

* Peripheral neurotoxicity > NCI grade 2
* Sever infection
* Previous history with chemotherapy or radiation therapy
* Pleural effusion, pericardial effusion, and ascites which could cause dyspnea > NCI grade 2
* Paraaortic lymph node metastasis
* Allergy with platinum
* Previous history of atrial or ventricular arrhythmia or congestive heart failure
* Uncontrolled infection, diabetes mellitus, hypertension, ischemic heart disease, myocardiac infarct within 6 months
* Severe disease such as acute or chronic renal failure and acute cerebral infarct, cerebral hemorrhage, recurrent hepatitis, liver cirrhosis, unknown fever above 39 degrees centigrade

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Care clinic
Sampling Method: Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2012-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Weon Kim, Professor, Study Director — Seoul National University Hospital; Seung Su Han, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea